CLINICAL TRIAL: NCT02549105
Title: A Comparison Between Lidocaine-Prilocaine Cream (EMLA) Application And Wound Infiltration With Lidocaine For Post Caesarean Section Pain Relief : A Randomized Controlled Trial
Brief Title: Lidocaine-Prilocaine Cream (EMLA) Topical Application Versus Wound Infiltration With Lidocaine After Cesarean Section
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Principal Investigator, HANY AYAD IBRAHIM, RESIDENT DOCTOR, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ain Shams MH
Record Dates: First submitted 2015-01-21; First posted 2015-09-15 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Post Operative Pain
Keywords: EMLA CREAM; LIDOCAINE INFILTERATION; PAIN RELIEF
MeSH Terms: conditions — Pain, Postoperative | interventions — Lidocaine, Prilocaine Drug Combination; Lidocaine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EMLA CREAM (Active Comparator): EMLA CREAM 5 mg TOPICAL APPLICATION FOR CS WOUND AND ASSESSMENT FOR POST OPERATIVE PAIN IN FIRST 6 HOURS
  Interventions: Drug: EMLA CREAM 5 mg
- LIDOCAINE INFILTERATION (Active Comparator): LIDOCAINE 1 % 20 ml INFILTERATION FOR WOUND AND ASSESSMENT OF POST OPERATIVE PAIN IN FIRST 6 HOURS
  Interventions: Drug: LIDOCAINE 1 %

INTERVENTIONS:
Drug: EMLA CREAM 5 mg — EMLA CREAM APPLICATION FOR WOUND AFTER CS
  Other Names: EMLA CREAM, PRILOCAIN 25 LIDOCAIN 25
  Arms: EMLA CREAM
Drug: LIDOCAINE 1 % — LIDOCAINE 1 % INFILTERATION FOR WOUND AND ASSESSMENT OF PAIN IN FIRST 6 HOURS
  Other Names: XYLOCAINE
  Arms: LIDOCAINE INFILTERATION

SUMMARY:
A Comparison Between Lidocaine-Prilocaine Cream (EMLA) Application And wound Infiltration with Lidocaine For Post Caesarean Section Pain Relief : A Randomized Controlled Trial.

DETAILED DESCRIPTION:
The purpose of this study is to compare the effectiveness of topically applied lidocaine-prilocaine (EMLA) cream with local anesthetic (lidocaine) infiltration on post-cesarean section pain.

Research Question:

Is lidocaine-prilocaine (EMLA) cream application effective as compared to local anesthetic (lidocaine) infiltration on post-caesarean section pain?

Research Hypothesis:

Lidocaine-prilocaine (EMLA) cream application is effective in post_caesarean section pain as compared to local anesthetic (lidocaine) infiltration.

Clinical Application :

Topical Lidocaine-prilocaine (EMLA) cream could be applied frequent times postoperatively, unlike infiltration with local anesthetic.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 40 years.
2. Patient American Society of Anesthesiologists physical status І or П.
3. Gestational age of pregnancy of 37w or more.
4. Patient have no previous section or have 1or 2 previous sections.
5. Patient having no medical disorders.
6. Patient with no obstetrical complications.

Exclusion Criteria:

1. age below18 or above 40.
2. Women American Society of Anesthesiologists physical status ш or more.
3. Women having more than 2 previous cesarean section.
4. Women receive cardio vascular drugs or having history of cardio vascular disease.
5. Women with Medical disorders with pregnancy as diabetes milletus.
6. Women having obstetrical complications as antepartum hemorrhage, pre-eclampsia or eclampsia.
7. Women having metabolic, hormonal, respiratory, renal and hepatic disease.
8. Women with any severe allergic condition or severe asthma.
9. Mental condition rendering the patients unable to understand the nature, scope and possible consequences of the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
TIME TO THE FIRST DOSE OF RESCUE ANALGESIC IN THE FIRST 6 HOURS | 6 H

SECONDARY OUTCOMES:
POSTOPERATIVE PAIN ACCORDING TO VAS | 24 H

CONTACTS AND LOCATIONS:
Overall Officials: MAGED R ABO SAEDA, MD, Principal Investigator — AIN SHAMS MATERNAL HOSPITAL
Locations (1):
- Ain Shams university Maternity hospital, Cairo, Abbasya, Egypt